CLINICAL TRIAL: NCT06615583
Title: A Novel Adaptive Anastomotic Technique for Left-sided Colonic and Rectal Resection: a Pilot, Single-center, Prospective, Case-series Study
Brief Title: A Novel Adaptive Anastomotic Technique for Left-sided Colonic Resection
Acronym: NOVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Carponovum AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR1-2024-102
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Colon Neoplasm
Keywords: Colorectal neoplasms; Colorectal anastomosis; Anastomotic leak; Surgical device
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Anastomotic Leak | interventions — Surgical Fixation Devices

STUDY DESIGN:
Intervention Model Description: Pilot, single-center, interventional, prospective, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- C-REX arm (Experimental): Patients will receive the C-REX device during sigmoid or high rectal resection. They will be instructed to follow a low residue diet and administered with a stool softener for five days after the surgical intervention. Approximately ten days after surgery, patients will release the study device and the anastomosis will be assessed with digital endoscopy.
  Interventions: Device: Surgical device

INTERVENTIONS:
Device: Surgical device — The C-REX device consists of an invasive surgical part, including two anastomotic rings, and surgical instruments for assisting the placement of the anastomotic ring to intestine. The rings are loosen from the inside of the intestinal wall and expelled with faeces per rectum once the anastomosis is healed in approximately ten days.

SUMMARY:
The goal of this pilot clinical trial is provide preminary evidence of the effectiveness of the C-REX device, developed by CarpoNovum AB, in preventing anastomotic leak and improving anastomosis healing after sigmoid or high rectal resection in patients with colon neoplasia. The primary aim of the study is to evaluate the rate of anastomotic leak in patients receiving the study device within 90 days from the surgical procedure.

DETAILED DESCRIPTION:
Despite technological advancements, the rate of anastomotic leak after left colon and high rectal resection remains high, around 20%. The device C-REX, developed by CarpoNovum, may help the anastomosis construction and promote its healing. This may lead to reduced anastomotic leak rate and severity. This study aims to collect preliminary evidence on the effectiveness of C-REX to develop a future larger multicentric trial. This pilot study will collect preliminary data on the rate and severity of 90-day anastomotic leak in patients receiving the C-REX device.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged equal or more than 18 years old, both men and women.
* Patients with a proven diagnosis of sigmoid colon or high rectal tumors requiring anterior rectal resection as procedure of choice (colorectal cancer or benign polyps), as confirmed by radiological and histological exams.
* Patient indicated to minimally invasive or open sigmoid or high rectal resection.

Exclusion Criteria:

* Patients with pre-existing health conditions requiring surgery, such as intestinal obstruction or perforation, local or systemic infections, peritonitis, or intestinal ischemia. Patients with intraoperative evidence of any of these conditions will be withdrawn from the study.
* Patients with preoperative evidence of distal metastasis. Patients with intraoperative evidence of distal metastasis or peritoneal carcinosis will be withdrawn from the study.
* Patients with documented intestinal or anal stenosis or other obstructions distal to the anastomosis. Patients with intraoperative evidence of intestinal or anal stenosis will be withdrawn from the study.
* Patients who received radiation therapy to organs in abdomen or pelvis unrelated to current colorectal condition.
* Patients who are unable or received contraindication for the preoperative mechanical preparation. Patients with a preoperative evidence or suspicion of incomplete colon cleansing will be withdrawn from the study.
* Patients indicated to defunctioning stoma. Patients requiring diverting stoma as for intraoperative indication will be withdrawn from the study.
* Patients with an anastomosis in rectum below the peritoneal reflection and/or another procedure of choice than high anterior resection.
* Any condition that, in the opinion of the investigator, may interfere with the study conduction. In particular, any condition which can cause significant alteration of colonic wall thickness such as chronic and repeated infection which may impair the use of C-REX.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak rate | 90 days after surgery
  Rate of radiologically confirmed anastomotic leaks and their severity according to the International Study Group of Rectal Cancer (ISGR) grade

SECONDARY OUTCOMES:
Intraoperative anastomotic failures | Intraoperative
  Rate of intraoperative anastomotic construction failures, as confirmed by positive air leak test, reverse air leak test, or C-REX integrity pressure test after anastomosis construction
Time of anastomosis construction | Intraoperative
  Median time (in minutes) required to construct the anastomosis using the C-REX device
Time of C-REX evacuation | Ten days after surgery
  Median time required to evacuate the anastomotic ring of the C-REX device, in days
Anastomosis stenosis incidence rate | 90 days after surgery
  Incidence rate of anastomotic stenosis, as confirmed by digital endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, M.D., Ph.D., Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No
As for local Standard Operative Procedure, IPD will be stored in a public repository with appropriate embargo. Aggregate or psuedo-anonymized data will be shared only upon reasonable request